CLINICAL TRIAL: NCT02569853
Title: DFN-11 Injection in Episodic Migraine With or Without Aura
Acronym: RESTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFN-11-CD-004
Record Dates: First submitted 2015-10-01; First posted 2015-10-07 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Episodic Migraine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFN-11 (Experimental): DFN-11 active injection upon occurrence of migraine
  Interventions: Drug: DFN-11
- Placebo (Placebo Comparator): Placebo injection upon occurrence of migraine
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DFN-11
  Arms: DFN-11
Other: Placebo
  Arms: Placebo

SUMMARY:
Safety and Efficacy of DFN-11 in patients with episodic migraines with or without aura.

ELIGIBILITY:
Inclusion Criteria:

1. If female, a subject must have a negative serum pregnancy test at screening, does not plan to become pregnant during the study, and is not lactating
2. If female, a subject also must have a negative urine pregnancy test at all subsequent study visits after the Screening Visit, and agree to practice a reliable form of contraception or abstinence during the study. Acceptable forms of contraception include implants, injectables, combined oral contraceptives, an intrauterine device, a vasectomized partner, an exclusively female partner, and double-barrier methods.
3. If male (with female partner), a subject must agree to practice a reliable form of contraception or abstinence during the study.
4. A history of episodic migraine who experience 2 to 6 migraine attacks a month for at least the past 12 months with no more than 14 migraine headache days per month, and with 48 hours of headache free time between migraine headaches
5. Have migraine with or without aura; if with aura, the aura cannot last longer than 60 minutes

Exclusion Criteria:

1. Minors, even if they are in specified study age range
2. Medication overuse headache as defined by ICHD II:

   * Opioids ≥ 10 days a month during the 90 days prior to screening
   * Combination medications (e.g., Fiorinal®) ≥ 10 days a month during the 90 days prior to screening
   * Nonsteroidal anti-inflammatory drugs (NSAIDs) or other simple medications > 14 days a month during the 90 days prior to screening
   * Triptans or ergots ≥ 10 days a month during the 90 days prior to screening
3. Subjects treated with onabotulinumtoxin A (Botox®) or other botulinum toxin treatment; or history of receiving such treatment during the 180 days prior to screening
4. On unstable dosages of migraine prophylactic medications during the 30 days prior to and through screening
5. Taking mini-prophylaxis for menstrual migraine
6. Subjects with hemiplegic or basilar migraine or other forms of neurologically complicated migraine
7. Subjects who have prolonged aura (i.e., more than 1 hour)
8. Cerebrovascular disease including but not limited to a history of stroke or transient ischemic attack (TIA)
9. A history of migralepsy (seizure following a migraine) or a concurrent diagnosis of seizure disorder
10. Subjects who cannot differentiate between a migraine headache and tension-type or cluster headache or other types of headache
11. Subjects with a history of more than occasional (based on Investigator's judgment) tension-type headache (distinct from migraine headache days count).
12. Subjects with a history of cluster headaches
13. Subjects with the diagnosis of "probable migraine" (ICHD II)
14. Ischemic coronary artery disease (CAD): including but not limited to angina pectoris, history of myocardial infarction or documented silent ischemia or coronary artery vasospasm, including Prinzmetal's angina
15. Subjects with Wolff-Parkinson-White syndrome or arrhythmias associated with other cardiac accessory conduction pathway disorders
16. Subjects with a history of congenital heart disease
17. A history of uncontrolled hypertension or screening systolic/diastolic > 140/90 mmHg
18. Have peripheral vascular disease including but not limited to ischemic bowel disease (IBD) and Raynaud's disease.
19. Any abnormal physiology and/or pathology which, in the opinion of the Investigator or Sponsor, which would be contraindicated for study participation and would not allow the objectives of the study to be met
20. Subjects who show any clinical laboratory or electrocardiogram (ECG) abnormality that in the opinion of the Investigator would endanger the subject or interfere with the study conduct. If the results of the clinical laboratory or ECG are outside of normal reference range the subject may still be enrolled but only if these findings are determined to be not clinically significant by the Investigator. This determination must be recorded in the subject's source document prior to enrolment.
21. Fridericia's corrected QT (QTcF) interval greater than 450 msec
22. Severe renal impairment (creatinine > 2 mg/dl)
23. Serum total bilirubin > 2.0 mg/dL
24. Serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase > 2.5 times the upper limit of normal
25. Subjects with uncontrolled diabetes mellitus, or a glycosylated hemoglobin (HbA1c) > 7.0%, or with diabetes mellitus requiring insulin
26. A history of alcohol or substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Edition V (DSM-V) (including marijuana) within 1 year prior to screening
27. Current treatment with antipsychotics or use of antipsychotics within 30 days of screening
28. A history of or current neurological or psychiatric impairment, including but not limited to psychosis, current major depression, bipolar disorder or cognitive dysfunction that, in the opinion of the Investigator, would compromise data collection
29. Subjects who have received treatment with an investigational drug or device within 30 days of the screening visit or participated in a central nervous system clinical trial in the 3 months prior to screening
30. Subjects with any other medical condition that, in the judgment of the Investigator and/or Medical Monitor, would confound the objectives of the study (e.g., positive screening test for human immunodeficiency virus [HIV], hepatitis B surface antigen positive or hepatitis C positive, a known history of systemic lupus erythematosis)
31. Subjects who plan to donate blood, sperm, or oocytes during the study and for 30 days after the last dose of study medication
32. Subjects who are employees or immediate relatives of the employees of the Sponsor, any of its affiliates or partners, or of the study center

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2018-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Dr. Reddy's Investigational Site #18, Santa Monica, California
  - Dr. Reddy's Investigational Site #24, Jacksonville, Florida
  - Dr. Reddy's Investigational Site #23, Maitland, Florida
  - Dr. Reddy's Investigational Site #27, Boise, Idaho
  - Dr. Reddy's Investigational Site #20, Watertown, Massachusetts
  - Dr. Reddy's Investigational Site #19, Ann Arbor, Michigan
  - Dr. Reddy's Investigational Site #13, Springfield, Missouri
  - Dr. Reddy's Investigational Site #12, Albuquerque, New Mexico
  - Dr. Reddy's Investigational Site #10, Williamsville, New York
  - Dr. Reddy's Investigational Site #26, Greensboro, North Carolina
  - Dr. Reddy's Investigational Site #15, Cleveland, Ohio
  - Dr. Reddy's Investigational Site #21, Mt. Pleasant, South Carolina
  - Dr. Reddy's Investigational Site #25, Memphis, Tennessee
  - Dr. Reddy's Investigational Site #14, Dallas, Texas
  - Dr. Reddy's Investigational Site #16, Hurst, Texas
  - Dr. Reddy's Investigational Site #17, West Jordan, Utah

REFERENCES:
- [Derived] Landy S, Munjal S, Brand-Schieber E, Rapoport AM. Efficacy and safety of DFN-11 (sumatriptan injection, 3 mg) in adults with episodic migraine: a multicenter, randomized, double-blind, placebo-controlled study. J Headache Pain. 2018 Aug 15;19(1):69. doi: 10.1186/s10194-018-0881-z. PMID 30112726
- [Derived] Landy S, Munjal S, Brand-Schieber E, Rapoport AM. Efficacy and safety of DFN-11 (sumatriptan injection, 3 mg) in adults with episodic migraine: an 8-week open-label extension study. J Headache Pain. 2018 Aug 15;19(1):70. doi: 10.1186/s10194-018-0882-y. PMID 30112725

RESULTS

PARTICIPANT FLOW:
Groups:
- DFN-11 - Double-Blind: DFN-11 active injection upon occurrence of migraine
  DFN-11
- Placebo - Double-Blind: Placebo injection upon occurrence of migraine
  Placebo
Period: Overall Study
Arm/Group | DFN-11 - Double-Blind | Placebo - Double-Blind
Started | 131 | 137
Completed | 111 | 123
Not Completed | 20 | 14
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Did not experience migraine attack | 10 | 7
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFN-11 - Double-blind | Placebo - Double-blind | Total
Number analyzed (Participants) | 131 | 137 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (12.47) | 40.2 (12.28) | 41.0 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 111 | 118 | 229
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 29 | 23 | 52
  White | 98 | 105 | 203
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 131 | 137 | 268

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects in the Double-blind Period Who Are Pain Free at 2 Hours After Dosing as Reported by the Subject in the eDiary
Time Frame: 2 hours
Population: Subjects analyzed had efficacy data at the time of specified assessment
Measure: Number; unit: Percentage of responders
Arm/Group | DFN-11 - Double-Blind | Placebo - Double-Blind
Number analyzed (Participants) | 104 | 104
Percentage of responders | 51.0 | 30.8

2. Secondary Outcome: The Percentage of Subjects in the Double-blind Period Who Are Pain Free at 1 Hour After Dosing as Reported by the Subject in the eDiary
Time Frame: 1 hour
Population: Subjects analyzed had efficacy data at the time of specified assessment
Measure: Number; unit: Percentage of responders
Groups:
- DFN-11: DFN-11 active injection upon occurrence of migraine
  DFN-11
- Placebo: Placebo injection upon occurrence of migraine
  Placebo
Arm/Group | DFN-11 | Placebo
Number analyzed (Participants) | 104 | 101
Percentage of responders | 34.6 | 19.8

ADVERSE EVENTS:
Time Frame: During the double-blind treatment period, treatment-emergent adverse events were collected for 5 days after each time a subject treated a migraine with the study drug (DFN-11 or placebo).
Arm/Group | DFN-11 - Double-blind | Placebo - Double-blind
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/137
Other Adverse Events (participants affected / at risk) | 37/131 | 16/137
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFN-11 - Double-blind (N=131) | Placebo - Double-blind (N=137)
Injection site reaction (General disorders) | 24 (29) | 14 (18)
Paraesthesia (General disorders) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT02569853/Prot_SAP_000.pdf